CLINICAL TRIAL: NCT05920564
Title: Efficacy of Upper Trapezius Stretching on Neck Pain, Range of Motion and Disability in Patients With Cervical Spondylosis: A Randomised Controlled Trial
Brief Title: Upper Trapezius Stretching in Patients With Cervical Spondylosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/7780002023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Upper fibers of trapezius stretching; Other: Standard care
- Control group (Active Comparator)
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Upper fibers of trapezius stretching — The Upper fibers of trapezius stretching intervention involves specific stretching exercises designed to target the upper fibers of the trapezius muscle. The stretching exercises will be performed under the guidance of a licensed physical therapist and will involve extending the neck while gently pulling the head downward to stretch the upper fibers of the trapezius muscle. The intervention is designed to improve neck range of motion, reduce pain intensity, and reduce disability in patients with cervical spondylosis. The duration and frequency of the stretching exercises will be standardized across participants, and adherence will be monitored throughout the study period.
  Arms: Intervention group
Other: Standard care — The Control Group in this study will receive standard care, including heat treatment and strengthening exercises, but will not receive the specific Upper fibers of trapezius stretching intervention that is being tested in the Treatment Group.

SUMMARY:
This study aims to investigate the effectiveness of upper trapezius stretching exercises on pain intensity, neck range of motion, and disability in patients with cervical spondylosis. Patients with diagnosed cervical spondylosis will be randomly assigned to either a study group performing upper trapezius stretches or a control group. Both groups will receive heat treatment and strengthening exercises. The study group will additionally perform specific upper trapezius stretching exercises. Outcomes measures will be assessed before and after 4 weeks of intervention and will include neck pain intensity, range of motion, and disability using the Neck Disability Index. The study hypothesizes that the study group will demonstrate greater improvements in pain, range of motion, and disability compared to the control group. The study findings could provide data to guide physical therapy management of cervical spondylosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cervical spondylosis confirmed by orthopedic specialist
* Presence of neck pain for at least 3 months
* willingness to participate in the study and comply with the intervention

Exclusion Criteria:

* Recent neck trauma or fractures (within 6 months)
* Previous neck surgery
* Concurrent medical conditions that could affect neck pain and range of motion (e.g. rheumatoid arthritis)
* Concurrent physical therapy or rehabilitation for neck or shoulder
* Use of corticosteroids within past 3 months
* Pregnancy or serious circulatory conditions (due to use of heat pack)
* Known hypersensitivity to heat or cold
* Cognitive impairment that could interfere with ability to understand and complete self-report questionnaires and comply with interventions

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-06-28 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Neck pain intensity | Changes in neck pain intensity at baseline and after 4 weeks of intervention and 3 months
  elf-reported pain intensity in the neck region using a numerical rating scale (NRS).
Changes in Neck range of motion | Changes in neck range of motion at baseline and after 4 weeks of intervention and 3 months
  Degree of neck flexion, extension, lateral flexion and rotation using a goniometer.

SECONDARY OUTCOMES:
Changes in Neck Disability Index | Changes in Neck Disability Index at baseline and after 4 weeks of intervention and 3 months
  Self-reported disability due to neck pain based on a 10-item questionnaire covering pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Scored from 0-50, higher scores indicate greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No